CLINICAL TRIAL: NCT00202033
Title: Impact of Self-Monitoring Blood Glucose Frequency on Glycemic Control in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01856-04-C
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes
Keywords: referred to; comprehensive; diabetes; education; program
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): self monitor blood glucose 3 times a day per usual diabetes class curriculum
  Interventions: Behavioral: frequency of self monitoring blood glucose
- 2 (Experimental): only self monitor blood glucose when fasting
  Interventions: Behavioral: frequency of self monitoring blood glucose
- 3 (Experimental): no self monitoring of blood glucose
  Interventions: Behavioral: frequency of self monitoring blood glucose

INTERVENTIONS:
Behavioral: frequency of self monitoring blood glucose — Evaluate the impact of self monitoring blood glucose frequency on glycemic control in patients with type 2 diabetes.

SUMMARY:
To determine if the frequency of blood glucose testing in patients with type 2 diabetes who are being treated with diet and exercise alone or diet and exercise plus oral agents will impact the HbA1c level.

DETAILED DESCRIPTION:
To determine the impact of SMBG frequency on blood glucose control in patients receiving systematic diabetes management education through Type 2 Diabetes BASICS at International Diabetes Center.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Treatment with diet and exercise alone or with the addition of 1 or 2 oral agents
* Enrolled in Type 2 BASICS program
* A1c between 7.0 and 11%, inclusive
* Able to understand spoken English

Exclusion Criteria:

* Insulin therapy
* Unable/unwilling to perform SMBG
* Participating in another research study
* Currently performing SMBG >3 times/week

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
HbA1c | 2 years

SECONDARY OUTCOMES:
blood glucose testing frequency | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bergenstal, MD, Principal Investigator — Park Nicollet Institute/International Diabetes Center
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States